CLINICAL TRIAL: NCT04519164
Title: Aldosterone, the Mineralocorticoid Receptor, and Cardiovascular Disease in Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Anand Vaidya, Associate Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P002311
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Syndrome; Hypertension; Overweight and Obesity
Keywords: aldosterone; mineralocorticoid receptor antagonist
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Overweight; Obesity | interventions — Eplerenone; Chlorthalidone; Potassium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive either eplerenone or chlorthalidone with potassium chloride
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: study medications will be blinded to the participant, investigator, outcomes assessors, and the care providers of the participants. Only the research pharmacists who prepare the study medications will be aware.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Eplerenone (Experimental): Participants will receive eplerenone, ranging from 25-100mg daily for one year.
  Interventions: Drug: Eplerenone
- Chlorthalidone with potassium chloride (Active Comparator): Participants will receive chlorthalidone (6.25-25mg daily for one year) along with potassium chloride (up to 20 mEq daily for one year)
  Interventions: Drug: Chlorthalidone with potassium chloride

INTERVENTIONS:
Drug: Eplerenone — mineralocorticoid receptor antagonist and potassium-sparing diuretic
  Other Names: Inspra
  Arms: Eplerenone
Drug: Chlorthalidone with potassium chloride — potassium-wasting diuretic with potassium chloride
  Other Names: hygroton
  Arms: Chlorthalidone with potassium chloride

SUMMARY:
This study will evaluate whether the mineralocorticoid receptor antagonist eplerenone, when compared to chlorthalidone plus potassium chloride, can improve cardiac MRI-derived myocardial perfusion reserve and fibrosis, independent of blood pressure, and proportionately to the severity of autonomous aldosterone production.

DETAILED DESCRIPTION:
Obesity is a dominant risk factor for the development of cardiovascular disease (CVD). The public health relevance of this relationship is underscored by the fact that 40% (93 million) of adult Americans are obese.

Activation of the mineralocorticoid receptor (MR) is a major mechanism implicated in the pathogenesis of obesity-associated CVD. MR activation causes vascular stiffness, inflammation, and fibrosis, and MR antagonists improve clinical outcomes in heart failure with reduced ejection fraction, especially in obesity. However, even in the absence of heart failure, multiple mechanisms of CVD in obesity are mediated by excessive activation of the MR. These mechanisms include: autonomous aldosterone production, increased cortisol action, high sympathetic nervous system activity, increased leptin, inflammation, and oxidative stress.

Autonomous aldosterone production is a highly prevalent and poorly recognized disorder that causes CVD independent of blood pressure (BP). Autonomous aldosterone production manifests across a wide severity spectrum, ranging from mild/subclinical (rarely recognized) to overt (primary aldosteronism). The investigators' work has characterized autonomous aldosterone production as a phenotype of non-physiologic, non-suppressible, and renin-independent aldosterone production that is highly prevalent in the general population of the U.S.A..

Autonomous aldosterone production and MR activation are especially enriched in obesity, particularly among obese/overweight individuals with hypertension and/or metabolic syndrome. Current treatment guidelines do not recommend the early use of MR antagonists in obesity or hypertension, thereby delaying or omitting a targeted therapy that may specifically mitigate the mechanism of CVD in this high-risk population.

The investigators have validated cardiac MRI methods to measure coronary microvascular function and myocardial fibrosis, both strong surrogates for CVD that correlate with aldosterone production and that improve with MR antagonist therapy.

Prospective studies to investigate the early mechanistic contribution of aldosterone-MR activation in the pathogenesis of CVD in obesity, and whether MR antagonists can prevent this, are lacking. Mechanistic studies, using innovative and robust intermediate phenotypes of clinical CVD outcomes in a cost-effective manner, could have a major public health impact by implicating a targeted medical therapy (MR antagonists) to prevent CVD in high-risk obesity (overweight/obese individuals with hypertension and/or metabolic syndrome).

HYPOTHESIS: MR antagonists in high-risk obesity improve cardiac MRI-derived myocardial perfusion reserve and fibrosis, independent of BP, and proportionately to the severity of autonomous aldosterone production.

STUDY DESIGN: This mechanistic study will investigate whether MR antagonist therapy in high-risk overweight or obese participants can be a targeted strategy to prevent CVD.

80 participants with overweight/obesity, untreated hypertension, and/or at least one other feature of the metabolic syndrome, will be enrolled. Participants will undergo a deep-phenotyping protocol to characterize aldosterone and cortisol physiology before randomization to eplerenone (25-100 mg/d) or chlorthalidone (6.25-25 mg/d + KCl 20 mEq/d) for one year. BP will be maintained in a target range to ensure outcomes are independent of BP control. Cardiac MRI-derived outcomes will be measured at baseline and after one year.

AIM 1: To investigate whether eplerenone therapy in high-risk obese/overweight participants, when compared to chlorthalidone + KCl, can improve coronary microvascular function independent of BP, as measured via stress cardiac MRI-derived myocardial perfusion reserve (a strong predictor for incident cardiovascular events and death that has been shown to improve with MR antagonist therapy).

AIM 2: To investigate whether eplerenone therapy in high-risk obese/overweight participants, when compared to chlorthalidone + KCl, can decrease myocardial fibrosis independent of BP, as measured via extracellular volume fraction on T1 mapping cardiac MRI (an established surrogate for myocardial fibrosis and inflammation that is also strongly associated with autonomous aldosterone production and mortality).

Exploratory Aims: To investigate whether the severity of autonomous aldosterone production is associated with cardiac MRI-derived outcomes and predicts the response to eplerenone therapy; and, to investigate whether eplerenone therapy can improve measures of cardiac fat content, arterial stiffness (via pulse-wave velocity), and inflammation (via inflammatory markers and adipocytokines), when compared to chlorthalidone + KCl.

IMPACT: Obesity/overweight status is enriched with autonomous aldosterone production and MR activation, mechanisms known to cause CVD. This study will investigate targeted mechanisms for the prevention of MR-mediated CVD in high-risk obesity using innovative physiologic phenotyping and surrogate imaging outcomes. This study will establish a mechanistic foundation for future outcome studies in obesity with incident CVD events.

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥ 30 with at least one of the following, or BMI ≥ 25 with at least two of the following:

   1. Untreated Hypertension: Stage I (BP 120-139/80-89 mmHg) or stage II (BP 140-159/90-99 mmHg).
   2. Treated Hypertension: On one anti-hypertensive medication with BP<140/90 mmHg and willing to undergo a 2-week washout of the medication before initiating eplerenone or chlorthalidone + KCl
   3. Dysglycemia: Impaired fasting plasma glucose (100-125 mg/dL) or glycated A1c 5.7-6.4%
   4. Dyslipidemia: Fasting triglyceride level > 150 mg/dL and HDL< 40 mg/dL in men or <50 mg/dL in women.
2. Age between 18 and 70 years old

Exclusion Criteria:

* Estimated glomerular filtration rate < 60 mL/min/1.73m2)
* Serum potassium > 5.2 mEq/L
* Known diagnosis or treatment for type 1 or type 2 diabetes
* Known history of CVD (myocardial infarction, heart failure, atrial fibrillation, or stroke)
* EKG with ischemic ST-segment or T-wave changes or Q waves in more than one territorial lead or a left bundle branch block
* Pregnancy (verified with a pregnancy test) or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Change in stress myocardial perfusion reserve on cardiac MRI | one year
  Change in myocardial perfusion

SECONDARY OUTCOMES:
Change in extracellular volume fraction on cardiac MRI | one year
  change in myocardial fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Anand Vaidya, MD, Principal Investigator — Brigham and Women's Hospital, Harvard Medical School
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No